CLINICAL TRIAL: NCT06003257
Title: Comparison Between Stainless-Steel, Zirconia and Fiberglass Crowns as Full Coverage Restoration for Deciduous Molars of Children
Brief Title: Comparison Between Stainless-Steel, Zirconia and Fiberglass Crowns for Deciduous Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 286/2020
Record Dates: First submitted 2023-07-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Caries of Infancy

STUDY DESIGN:
Intervention Model Description: Group I: comprise of 22 primary molars that will be subdivided into two subgroups:
  Subgroup IA: includes 11 primary molars will be restored by stainless steel crowns.
  Subgroup IB: includes 11 primary molars will be restored by zirconia crowns.
  Group II: comprise of 22 primary molars that will be subdivided into two subgroups:
  Subgroup IIA: includes 11 primary molars will be restored by stainless steel crowns.
  Subgroup IIB: includes 11 primary molars will be restored by fiberglass crowns.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- primary molars will be restored by stainless steel crowns (Active Comparator)
  Interventions: Other: stainless steel crown
- primary molars will be restored by zirconia crowns (Active Comparator)
  Interventions: Other: zirconia crown
- primary molars will be restored by fiberglass crowns. (Active Comparator)
  Interventions: Other: fiberglass crown

INTERVENTIONS:
Other: stainless steel crown — stainless steel full coverage crown for deciduous teeth
  Arms: primary molars will be restored by stainless steel crowns
Other: zirconia crown — zirconia full coverage crown for deciduous teeth
  Arms: primary molars will be restored by zirconia crowns
Other: fiberglass crown — fiberglass full coverage crown for deciduous teeth
  Arms: primary molars will be restored by fiberglass crowns.

SUMMARY:
The study will be divided into two parts: In vivo part and in vitro part.In vivo part: It will be a randomized clinical trial using split mouth technique on 44 primary molars in children aged from 4-8 years old selected from outpatient clinic of Department of Pediatric Dentistry, Faculty of Dentistry, Suez Canal University. The selected primary molars will be divided randomly into two main groups ,each group will be subdivided into two subgroups according to types of crowns that will be used as follows:- Group I:- comprise of 22 primary molars that will be subdivided into two subgroups, subgroup IA:-includes 11 primary molars will be restored by stainless steel crowns and subgroup IB:-includes 11 primary molars will be restored by zirconia crowns, Group II:- comprise of 22 primary molars that will be subdivided into two subgroups, subgroup IIA:-includes 11 primary molars will be restored by stainless steel crowns and subgroup IIB:-includes 11 primary molars will be restored by fiberglass crowns. The three types of crowns will be evaluated at the baseline once after cementation of the crowns and after one week,1 ,3,6,9 and 12 months follow up by using the following methods modified United States Public Health Service criteria, in terms of color match, marginal integrity, secondary caries and crown fracture, the gingival marginal status and parental satisfaction. In vitro part: It will be carried out on 30 mandibular primary molars, 15 mandibular first primary molars for microleakage test and 15 mandibular second primary molars for crown fracture resistance test for three crowns types.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial using split mouth technique on 44 primary molars in children aged from 4-8 years old selected from outpatient Clinic of Department of Pediatric Dentistry, Faculty of Dentistry, Suez Canal University after approval of Research Ethics Committee (REC) of the Faculty of Dentistry, Suez Canal University. The children participants and legal guardian of each participant will be assigned on informed consent of treatment procedures they will receive.

A total of 44 primary molars will be included in this study using split mouth technique to ensure equalizing variables for both groups.

The selected primary molars will be divided randomly into two main groups, each group will be subdivided into two subgroups according to types of crowns that will be used as follows: -

* Group I: comprise of 22 primary molars that will be subdivided into two subgroups:

  * Subgroup IA: includes 11 primary molars will be restored by stainless steel crowns.
  * Subgroup IB: includes 11 primary molars will be restored by zirconia crowns.
* Group II: comprise of 22 primary molars that will be subdivided into two subgroups:

  * Subgroup IIA: includes 11 primary molars will be restored by stainless steel crowns.
  * Subgroup IIB: includes 11 primary molars will be restored by fiberglass crowns.

II.4 Clinical Procedures:

* Eligibility criteria will be verified after the clinical and periapical radiographic examination.
* The selected primary molars will be anesthetized to reduce discomfort during preparation.
* Tooth preparation and crown cementation will be performed for each tooth according to the manufacture's instruction for each type of crowns.

II.5 Methods of evaluation:

The evaluation of each crown will be assessed at the baseline once after cementation and after one week,1, 3, 6,9 and 12 months follow up by using the following methods:

II.5.1 Modified United States Public Health Service (USPHS) criteria:

Modified United States Public Health Service (USPHS) criteria will be used in terms of marginal integrity, secondary caries, color match, and crown fracture

ELIGIBILITY:
Inclusion Criteria:

* 1. Apparently healthy children free from any systemic diseases. 2. Patient within the age group of 4 to 8 years old of both sexes. 3. Cooperative patient. 4. Patient with at least two bilateral primary molars indicated for full coverage as follows:

  1. Multi-surfaces caries more than two surfaces
  2. Pulp therapy treated primary molars
  3. Developmental defects on tooth surface
  4. Root resorption less than/ equal to1/3rd of root length 5. Parent willing to participate in the study.

Exclusion Criteria:

* Patient with primary molars have the following criteria:

  1. Acute infection
  2. Infra-occlusion
  3. Mobility
  4. Internal root resorption
  5. Exfoliation imminent

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
clinical performance " marginal integrity, color change, secondary caries and crown fractures" | immediately after cementation, after 1 month, 3 months, 6 months, 9 months and 12 months
  Modified United States Public Health Service (USPHS) criteria will be used in terms of marginal integrity, secondary caries, color match, and crown fracture

SECONDARY OUTCOMES:
Measuring of gingival marginal status | immediately after cementation, after 1 month, 3 months, 6 months, 9 months and 12 months
  The gingival marginal status will be assessed by the plaque index (PI) and gingival index where 0 normal gingiva and no plaque while 3 severe inflammation and abudance of soft matter within gingival pocket
Measuring of parental satisfaction | immediately after cementation, after 1 month, 3 months, 6 months, 9 months and 12 months
  Parental satisfaction will be evaluated on a five-point Likert scale, which responders specify their level of satisfaction. parents will ask to rate parameters such as the crown's shape, size, color, and their overall satisfaction by using Parental satisfactions questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No